CLINICAL TRIAL: NCT04742140
Title: Magnesium Sulphate Injection in Treatment of Myofascial Trigger Points in Masseter Muscle
Brief Title: Magnesium Sulphate Injection in Treatment of Myofascial Trigger Points
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, associate professor in oral & maxillofacial Surgery Department, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mg SO4 injections
Record Dates: First submitted 2021-01-30; First posted 2021-02-05 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: trigger point; masseter muscle; myofascial pain; magnesium sulphate
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group I (Active Comparator): each patient injected 0.5ml in each TrPs of saline by the same operator
  Interventions: Drug: Saline
- group II (Experimental): each patient injected 0.5ml in each TrPs of magnesium sulphate by the same operator
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — each patient injected 0.5ml in each TrPs of magnesium sulphate according to the treatment group by the same operator
  Other Names: Study
  Arms: group II
Drug: Saline — each patient injected 0.5ml in each TrPs of saline according to the treatment group by the same operator
  Other Names: Control
  Arms: group I

SUMMARY:
This is a prospective, single- center, randomized (1:1) clinical trial comparing the effectiveness of magnesium sulphate injections in treatment of myofascial trigger points in the masseter muscle versus the saline injection.

DETAILED DESCRIPTION:
The proposal presents the magnesium sulphate (MgSO4) as a possible injection treatment for TrPs. The MgSO4 prevents the release of pre-synaptic acetylcholine from neuromuscular and sympathetic junctions that could explain the ability of the MgSO4 to relax the muscle and reduce pain Specific aim: evaluate the effectiveness of magnesium sulphate injections in treatment of myofascial trigger points in the masseter muscle versus the saline injection.

Hypothesis: the injection of masseter muscle trigger points with magnesium sulphate is more effective than saline injection in pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of myofascial pain with a referral, based on the DC/TMD criteria
* the presence of one or more trigger points in the unilateral or bilateral masseter muscle
* no history of any invasive procedures in the related masseter muscle.

Exclusion Criteria:

* Factors that can cause pain in the orofacial region other than MTPs (decayed tooth, TMJ internal disorder).
* Any systemic disease that possibly affects the masticatory system such as rheumatoid arthritis and epilepsy
* pregnancy and lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
pain score | 6 months postoperative
  pain score measured on a 10-point visual analogue scale (VAS), the 0 indicating no pain and 10 indicating the worst pain ever.

SECONDARY OUTCOMES:
quality-of-life in an Oral Health Impact Profile questionnaire (OHIP-14) | six months postoperative
  OHIP-14 is used to measure patients' self-reported discomfort, disability, and functional limitation due to oral conditions with scores ranging from 0 to 56 (with 56 representing a subject answering ''very often'' to all 14 items)

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Mohamed, phd, Principal Investigator — Fayoum University
Locations (1):
- Faculty of Dentistry, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yilmaz O, Sivrikaya EC, Taskesen F, Pirpir C, Ciftci S. Comparison of the Efficacy of Botulinum Toxin, Local Anesthesia, and Platelet-Rich Plasma Injections in Patients With Myofascial Trigger Points in the Masseter Muscle. J Oral Maxillofac Surg. 2021 Jan;79(1):88.e1-88.e9. doi: 10.1016/j.joms.2020.09.013. Epub 2020 Sep 14. PMID 33045182
- [Background] Yousef AA, Al-deeb AE. A double-blinded randomised controlled study of the value of sequential intravenous and oral magnesium therapy in patients with chronic low back pain with a neuropathic component. Anaesthesia. 2013 Mar;68(3):260-6. doi: 10.1111/anae.12107. Epub 2012 Dec 17. PMID 23384256
- [Background] Sakalys D, Rokicki JP, Januzis G, Kubilius R. Plasma rich in growth factors injection effectiveness for myofascial pain treatment in masticatory muscles. Randomised controlled trial. J Oral Rehabil. 2020 Jul;47(7):796-801. doi: 10.1111/joor.12973. Epub 2020 Apr 21. PMID 32271467
- [Derived] Refahee SM, Mahrous AI, Shabaan AA. Clinical efficacy of magnesium sulfate injection in the treatment of masseter muscle trigger points: a randomized clinical study. BMC Oral Health. 2022 Sep 19;22(1):408. doi: 10.1186/s12903-022-02452-3. PMID 36123724